CLINICAL TRIAL: NCT03695939
Title: An Open-label Phase 1/2 Study to Evaluate the Safety, Tolerability, and Efficacy of realSKIN® (Skin Xenotransplant) for Complete Closure of Severe and Extensive Deep-Partial and Full-Thickness Burn Wounds
Brief Title: Evaluation of Safety and Efficacy of realSKIN® (Skin Xenotransplant) for Complete Closure of Severe Burn Wounds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XenoTherapeutics, Inc. (Other)
Collaborators: Massachusetts General Hospital (Other); Joseph M. Still Research Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001839
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-12

CONDITIONS: Deep Full-thickness Burn Injury (Disorder)
Keywords: xenotransplant; skin; burns; temporary; allograft; porcine; closure; dressing; live biotherapeutic; xenograft; pig; genetically engineered; alpha-Gal; GalT-KO
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2, Open-label, Multi-center, Clinical Trial to evaluate the safety, tolerability, and efficacy of realSKIN® to provide complete wound closure of severe and extensive deep-partial or full-thickness burn wounds. Approximately 25 total subjects will be enrolled. The designated realSKIN® product size will be placed on the burn wound following wound site preparation, including necessary debridement and tangential excision as determined by burn surgeon and secured in place via suturing or stapling. The remaining burn wound will be covered with human cadaver allograft and treated according to local standard of care with care to avoid any overlap or significant contact of the two temporary wound dressings. The Investigator will assess the wounds and identify the matched pair of burn sites then the treatments will be randomly assigned to the sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment: realSKIN (skin xenotransplant) (Experimental): In the experimental arm, patients are treated with the investigational drug, realSKIN®, in a side-by-side comparison to the active comparator, thus, each patient serves as their own control. The designated realSKIN® product size will be placed on the burn wound and secured in place via suturing or stapling. The Investigator will assess the wounds and identify the matched pair of burn sites then the treatments will be randomly assigned to the sites.
  Interventions: Biological: realSKIN (skin xenotransplant)
- Active Comparator: Human Allograft Skin (Active Comparator): In the active comparator arm, patients are treated with human cadaver allograft, in a side-by-side comparison to the investigational drug, thus, each patient serves as their own control.
  The allograft active comparator will be placed adjacently to the investigational drug, in the same anatomical location, on wound sites following debridement and secured via suture or staples. All other treatment aspects were consistent with the standard of care. The Investigator will assess the wounds and identify the matched pair of burn sites then the treatments will be randomly assigned to the sites.
  Interventions: Biological: Human Cadaver Allograft

INTERVENTIONS:
Biological: realSKIN (skin xenotransplant) — 3+3 Dose-escalation Study Design; 2 dosage strengths will be utilized during this Phase 1/2 Trial; an expansion cohort (9 patients) receive the highest dose.
  Arms: Experimental Treatment: realSKIN (skin xenotransplant)
Biological: Human Cadaver Allograft — HCA is used as a temporary wound dressing between debridement and definitive closure in many well-resourced contexts.
  Other Names: Human Allograft Skin; HCA
  Arms: Active Comparator: Human Allograft Skin

SUMMARY:
This is a Phase 1/2, Open-label, Multi-center, Clinical Trial to evaluate the safety, tolerability, and efficacy of realSKIN® to provide complete wound closure of severe and extensive deep-partial and full-thickness burn wounds.

Approximately 25 total subjects will be enrolled. Subjects who meet eligibility criteria and provide written informed consent will receive realSKIN® placement at a single burn wound site. The designated realSKIN® product size will be placed on the burn wound following wound site preparation, including necessary debridement and tangential excision as determined by burn surgeon and secured in place via suturing or stapling. The remaining burn wound will be covered with human cadaver allograft and treated according to local standard of care with care to avoid any overlap or significant contact of the two temporary wound dressings. The Investigator will assess the wounds and identify the matched pair of burn sites then the treatments will be randomly assigned to the sites.

realSKIN® will remain in place until intentional removal per Investigator's direction consistent with subject's overall clinical course, or if it is deemed to no longer provide effective wound closure and barrier function to the wound bed. The Investigator will follow local standard of care relevant to wound care and dressing changes while the realSKIN® is in place. Standard of care burn management will be provided by the Investigator.

Routine vital sign assessments, photography, laboratory tests (hematology, chemistry, and urinalysis), physical exams, and adverse event monitoring will occur while realSKIN® is in place and for up to 1 year following initial placement. Subjects will be monitored via a passive and active screening program using blood samples collected at time points throughout the study period, as adapted from FDA Guidance for Industry.

The risk of transmission of infectious disease is expected to be extremely low and while limited human trial data are available there have been no reports of transmission of porcine microorganisms to humans, and to date, there have been no adverse events (AEs) related to the use of realSKIN® observed or reported, and independent analysis of PERV data and medical records by the Safety Review Committee has indicated no evidence of zoonotic transmission in this trial.

DETAILED DESCRIPTION:
Product Name: realSKIN®

Chemical Name: alpha-1,3-galactosyltransferase knock-out (GalT-KO) porcine (Sus scrofa) epidermal and dermal layers.

Chemical Structure: realSKIN® a biologically active, split-thickness, xenotransplantation skin product. realSKIN® is derived from specialized, genetically engineered (alpha 1,3 galactosyltransferase knockout [GalT-KO]), Designated Pathogen Free (DPF), porcine donors, containing vital, metabolically active (i.e., non-terminally sterilized) porcine cells within the dermal and epidermal tissue layers.

Proposed Indication: realSKIN is indicated for the treatment of mixed-depth, full-thickness burn wounds requiring hospitalization, surgical excision, and skin grafting.

Drug Type: realSKIN® is classified as a Live Biotherapeutic Product (LBP). (Guidance to Industry, Early Clinical Trials with Live Biotherapeutic Products, Section 1.b.)

Active Ingredient: Live (i.e. non-terminally sterilized) porcine cells, including endothelial cells of intact vasculature and those comprising the dermal and epidermal tissue layers

Product Structure: realSKIN® has an approximate thickness of 0.022 inches (0.55mm) and is currently provided in one investigational size: approximately 5x15 cm2 (22.5g/75 cm2).

Formulation: Each lot or releasable batch of realSKIN® is derived from a single source animal and each batch is independently processed and tested for various adventitious agents, histology, morphology, sterility, and purity.

Route of Administration: Surgical engraftment, via sutures or staples

Dosing Regimen: A single topical application of realSKIN has an approximate size of 150 cm2, with dimensions of 5 cm x 15 cm, meshed in a 2:1 ratio, and has an approximate thickness of 0.022 inches (0.55 mm).

realSKIN is intended for a one-time, topical application to a surgically prepared wound bed via sutures or staples and may be trimmed to fit the shape and size of the actual wound area. realSKIN can be used in the treatment of an overall injury size of up to 30% TBSA burn injury.

Drug's Mechanism of Action: realSKIN is intended for topical use directly on debrided, severe and extensive, mixed-depth and full-thickness burn wounds to provide complete and durable wound closure.

As a living skin transplant, realSKIN forms microvascular connections with host vessels in the burn wound bed which leads to wound closure. realSKIN replaces elements of whole, living skin that are analogous and functionally equivalent to those found in healthy human skin. realSKIN does not remain permanently engrafted but is replaced by the patient's own cells over time.

This mechanism of action distinguishes realSKIN from traditional xenograft products which are terminally sterilized, rendering the cells inactive, limiting their therapeutic capability to effect complete and durable wound closure.

Drug Packaging: Each realSKIN® product is individually packaged in a clear plastic, externally threaded, 10-ml polypropylene vial with threaded seal-cap, stored on a rolled, sterile nylon mesh backing on the dermal-side of the realSKIN® product that serves to support and protect the graft during processing and transport. Within this container, each realSKIN® product is individually immersed in 7-ml of sterile cryoprotective medium with 5% dimethyl sulfoxide (DMSO) (CryoStor CS5, BioLifeSolutions). Source animal serum is NOT included or used in this process. The contents are cryopreserved via controlled rate, phase freezer and stored at -80o C until use. All packaging materials are removed prior to the surgical procedure and dressing placement.

ELIGIBILITY:
Inclusion Criteria:

1. The subject provides written informed consent to participate in this study
2. Males or females age greater than 18 years old
3. Females must have a negative serum pregnancy test at Screening and at Baseline and must not be nursing
4. Male and female subjects must agree to use a protocol-approved method of contraception for a minimum of 3 months following Xeno-Skin® placement, which includes a barrier method plus one or more of the following:

   1. Hormonal contraceptives (e.g., birth control pills, skin patches, vaginal rings, and the Depo- Provera shot)
   2. Intrauterine device (IUD)
   3. Male or female condoms with spermicide
   4. Diaphragm with spermicide
   5. Permanent tubal occlusive birth control system
5. Total Body Surface Area (TBSA) <30%, to include deep-partial thickness or full-thickness burn wounds
6. Burn injuries would otherwise require debridement and tangential excision
7. Burn injury requiring temporary grafting with human cadaver allograft skin, based on clinical judgment prior to definitive wound closure via autologous grafting
8. Sufficient area of burn wound for Xeno-Skin® placement and not located on face or hands or having an engraftment site centered on high-impact areas such as joints, weight-bearing areas (e.g. soles of feet), or the inguinal region, per Investigator's judgment

Exclusion Criteria:

1. Pregnant or lactating women
2. Documented history of infection with human immunodeficiency virus (HIV) or other condition(s) that in the opinion of the Investigator may compromise patient safety or study objectives
3. Immunosuppressive medication regimens e.g. antineoplastics, high dose steroids (> 10 mg prednisone/day), TNF alpha inhibitors, calcineurin inhibitors (cyclosporine, tacrolimus), anti-proliferative agents, and other immunomodulators
4. Known allergy to penicillins (such as ampicillin), ceftazidime or aztreonam, glycopeptide antibiotics (such as vancomycin) or amphotericin B
5. Active malignancy, including those requiring surgery, chemotherapy, and/or radiation in the past 5 years. Non-metastatic basal or squamous cell carcinoma of the skin and cervical carcinoma in situ are allowed
6. Use of any experimental or investigational drugs within 30 days prior to placement of Xeno-Skin®
7. Previously received a porcine or other xenogeneic tissue product, including but not limited to: glutaraldehyde fixed porcine or bovine bioprosthetic heart valve replacements and glutaraldehyde fixed porcine dermal matrix (e.g., EZ Derm)
8. BMI > 40 kg/m2
9. HbA1c ≥ 7.0%
10. Treatment with systemic corticosteroids within 30 days before screening (not including inhaled steroids)
11. Electrical, chemical, or radiation burns
12. History of chronic end stage renal disease defined as an MDRD CrCl < 15 mL/min, or receiving chronic dialysis
13. History of chronic liver disease or cirrhosis (Child-Pugh Score C). Evidence of acute or chronic hepatitis B infection based on documented HBV serology testing
14. Known documented history of Hepatitis B, Hepatitis C, Treponema pallidum, Cytomegalovirus, herpes or varicella zoster Note: Successfully treated hepatitis C patients without evidence of end stage liver disease is allowed. If HCV antibody reactive, then HCV RNA must be undetectable.
15. Recent (within 3 months prior to study enrollment) MI, unstable angina leading to hospitalization, uncontrolled, CABG, PCI, carotid surgery or stenting, cerebrovascular accident, transient ischemic attack (TIA), endovascular procedure or surgical intervention for peripheral vascular disease or plans to undergo a major surgical or interventional procedure (eg, PCI, CABG, carotid or peripheral revascularization)
16. Presence of venous or arterial vascular disorder directly affecting the area of burn wound
17. Pre-existing haemolytic anemia
18. Chronic malnourishment as determined by Investigator
19. Significant pulmonary compromise
20. Systemic anticoagulation at the time of treatment or INR > 2
21. Documented evidence of wound infection at Screening or Baseline
22. Evidence of sepsis and/or end organ damage
23. Acute lung injury
24. Life expectancy of less than 180 days
25. Subject who is unable to self-consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Temporary Wound Closure | Prior to autograft placement (within 14 days)
  To assess the capability of realSKIN® to improve wound healing by providing supportive care until definitive closure can be accomplished by functioning as a barrier, much like human skin, as compared to similar wound site(s) treated with human cadaver allograft (HCA).
Long-term Safety and Tolerability | Prior to autograft placement (continued follow up through 6 months)
  To further demonstrate the long-term safety and tolerability of realSKIN®, to include evidence that Xeno-Skin® does not significantly impede wound healing.

SECONDARY OUTCOMES:
Definitive Wound Closure | Post autograft placement (continued follow up through 1 year)
  To assess the quality of healing, to include scarring, contour and feel of healed skin, or normalization of skin markings or pigmentation, at wound treatment sites that received temporary closure with realSKIN®, as compared to that of wound treatment site(s) that received temporary closure with human cadaver allograft (HCA).
Improved Wound Healing | Post autograft placement (continued follow up through 1 year)
  To assess the capability of realSKIN® to improve wound healing by providing supportive care until definitive closure can be accomplished by functioning as a barrier, much like human skin, as compared to similar wound site(s) treated with human cadaver allograft (HCA).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Goverman, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - JMS Burn Center at Doctors Hospital, Augusta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albritton A, Leonard DA, Leto Barone A, Keegan J, Mallard C, Sachs DH, Kurtz JM, Cetrulo CL Jr. Lack of cross-sensitization between alpha-1,3-galactosyltransferase knockout porcine and allogeneic skin grafts permits serial grafting. Transplantation. 2014 Jun 27;97(12):1209-15. doi: 10.1097/TP.0000000000000093. PMID 24798308
- [Background] Bruccoleri RE, Matthew MK, Schulz JT. Methods in obtaining split-thickness skin grafts from skin reduction surgery specimens. Springerplus. 2016 May 25;5(1):690. doi: 10.1186/s40064-016-2330-2. eCollection 2016. PMID 27350924
- [Background] Burd A, Chiu T. Allogenic skin in the treatment of burns. Clin Dermatol. 2005 Jul-Aug;23(4):376-87. doi: 10.1016/j.clindermatol.2004.07.019. PMID 16023933
- [Background] Denner J. Paving the Path toward Porcine Organs for Transplantation. N Engl J Med. 2017 Nov 9;377(19):1891-1893. doi: 10.1056/NEJMcibr1710853. No abstract available. PMID 29117497
- [Background] Deschamps JY, Roux FA, Sai P, Gouin E. History of xenotransplantation. Xenotransplantation. 2005 Mar;12(2):91-109. doi: 10.1111/j.1399-3089.2004.00199.x. PMID 15693840
- [Background] Ericsson TA, Takeuchi Y, Templin C, Quinn G, Farhadian SF, Wood JC, Oldmixon BA, Suling KM, Ishii JK, Kitagawa Y, Miyazawa T, Salomon DR, Weiss RA, Patience C. Identification of receptors for pig endogenous retrovirus. Proc Natl Acad Sci U S A. 2003 May 27;100(11):6759-64. doi: 10.1073/pnas.1138025100. Epub 2003 May 9. PMID 12740431
- [Background] Fishman JA. Screening of source animals and clinical monitoring for xenotransplantation. Xenotransplantation. 2007, 349-352.
- [Background] Fishman JA, Scobie L, Takeuchi Y. Xenotransplantation-associated infectious risk: a WHO consultation. Xenotransplantation. 2012 Mar-Apr;19(2):72-81. doi: 10.1111/j.1399-3089.2012.00693.x. PMID 22497509
- [Background] Godehardt AW, Rodrigues Costa M, Tonjes RR. Review on porcine endogenous retrovirus detection assays--impact on quality and safety of xenotransplants. Xenotransplantation. 2015 Mar-Apr;22(2):95-101. doi: 10.1111/xen.12154. Epub 2015 Jan 31. PMID 25641488
- [Background] Herndon DN. Total Burn Care, Expert Consult - Online. Elsevier Health Sciences; 2012.
- [Background] Johnson RM, Richard R. Partial-thickness burns: identification and management. Adv Skin Wound Care. 2003 Jul-Aug;16(4):178-87; quiz 188-9. doi: 10.1097/00129334-200307000-00010. PMID 12897674
- [Background] Kitala D, Kawecki M, Klama-Baryla A, Labus W, Kraut M, Glik J, Ryszkiel I, Kawecki MP, Nowak M. Allogeneic vs. Autologous Skin Grafts in the Therapy of Patients with Burn Injuries: A Restrospective, Open-label Clinical Study with Pair Matching. Adv Clin Exp Med. 2016 Sep-Oct;25(5):923-929. doi: 10.17219/acem/61961. PMID 28028957
- [Background] Leonard DA, Mallard C, Albritton A, Torabi R, Mastroianni M, Sachs DH, Kurtz JM, Cetrulo CL Jr. Skin grafts from genetically modified alpha-1,3-galactosyltransferase knockout miniature swine: A functional equivalent to allografts. Burns. 2017 Dec;43(8):1717-1724. doi: 10.1016/j.burns.2017.04.026. Epub 2017 Jun 8. PMID 28602591
- [Background] Leto Barone AA, Mastroianni M, Farkash EA, Mallard C, Albritton A, Torabi R, Leonard DA, Kurtz JM, Sachs DH, Cetrulo CL Jr. Genetically modified porcine split-thickness skin grafts as an alternative to allograft for provision of temporary wound coverage: preliminary characterization. Burns. 2015 May;41(3):565-74. doi: 10.1016/j.burns.2014.09.003. Epub 2014 Oct 16. PMID 25406888
- [Background] Organ Procurement and Transplantation Network. (n.d.). Retrieved May 01, 2017, from https://optn.transplant.hrsa.gov/
- [Background] Martin SI, Wilkinson R, Fishman JA. Genomic presence of recombinant porcine endogenous retrovirus in transmitting miniature swine. Virol J. 2006 Nov 2;3:91. doi: 10.1186/1743-422X-3-91. PMID 17081300
- [Background] Meije Y, Tonjes RR, Fishman JA. Retroviral restriction factors and infectious risk in xenotransplantation. Am J Transplant. 2010 Jul;10(7):1511-6. doi: 10.1111/j.1600-6143.2010.03146.x. PMID 20642677
- [Background] Morozov VA, Wynyard S, Matsumoto S, Abalovich A, Denner J, Elliott R. No PERV transmission during a clinical trial of pig islet cell transplantation. Virus Res. 2017 Jan 2;227:34-40. doi: 10.1016/j.virusres.2016.08.012. Epub 2016 Sep 24. PMID 27677465
- [Background] Paradis K, Langford G, Long Z, Heneine W, Sandstrom P, Switzer WM, Chapman LE, Lockey C, Onions D, Otto E. Search for cross-species transmission of porcine endogenous retrovirus in patients treated with living pig tissue. The XEN 111 Study Group. Science. 1999 Aug 20;285(5431):1236-41. doi: 10.1126/science.285.5431.1236. PMID 10455044
- [Background] Patience C, Takeuchi Y, Weiss RA. Infection of human cells by an endogenous retrovirus of pigs. Nat Med. 1997 Mar;3(3):282-6. doi: 10.1038/nm0397-282. PMID 9055854
- [Background] Sachs DH. The lure of transplantation. Clin Transpl. 2008:287-305. No abstract available. PMID 19708462
- [Background] Schaffer A. Cadaver Skin Fills the Gap in Burn Cases. New York Times. May 2, 2006.
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Sheridan RL, Tompkins RG. Skin substitutes in burns. Burns. 1999 Mar;25(2):97-103. doi: 10.1016/s0305-4179(98)00176-4. No abstract available. PMID 10208382
- [Background] Shi M, Wang X, Okamoto M, Takao S, Baba M. Inhibition of porcine endogenous retrovirus (PERV) replication by HIV-1 gene expression inhibitors. Antiviral Res. 2009 Aug;83(2):201-4. doi: 10.1016/j.antiviral.2009.04.011. Epub 2009 May 3. PMID 19414036
- [Background] Thorton JF and Gosman AA. Skin Grafts and Skin Substitutes. Baylor University Medical Center. 2004 10(1): 2-78
- [Background] Weiner J, Yamada K, Ishikawa Y, Moran S, Etter J, Shimizu A, Smith RN, Sachs DH. Prolonged survival of GalT-KO swine skin on baboons. Xenotransplantation. 2010 Mar-Apr;17(2):147-52. doi: 10.1111/j.1399-3089.2010.00576.x. PMID 20522247
- [Background] Wilhelm M, Fishman JA, Pontikis R, Aubertin AM, Wilhelm FX. Susceptibility of recombinant porcine endogenous retrovirus reverse transcriptase to nucleoside and non-nucleoside inhibitors. Cell Mol Life Sci. 2002 Dec;59(12):2184-90. doi: 10.1007/s000180200017. PMID 12568344
- [Background] Wood JC, Quinn G, Suling KM, Oldmixon BA, Van Tine BA, Cina R, Arn S, Huang CA, Scobie L, Onions DE, Sachs DH, Schuurman HJ, Fishman JA, Patience C. Identification of exogenous forms of human-tropic porcine endogenous retrovirus in miniature Swine. J Virol. 2004 Mar;78(5):2494-501. doi: 10.1128/jvi.78.5.2494-2501.2004. PMID 14963150
- [Background] World Health Organization Burn Fact Sheet. http://www.who.int/en/news-room/fact-sheets/detail/burns. March 6, 2018.
- [Background] Wynyard S, Nathu D, Garkavenko O, Denner J, Elliott R. Microbiological safety of the first clinical pig islet xenotransplantation trial in New Zealand. Xenotransplantation. 2014 Jul-Aug;21(4):309-23. doi: 10.1111/xen.12102. Epub 2014 May 7. PMID 24801820
- [Background] Yue S, Zhang Y, Gao Y. A study on the susceptibility of allogeneic human hepatocytes to porcine endogenous retrovirus. Eur Rev Med Pharmacol Sci. 2015 Sep;19(18):3486-91. PMID 26439047
- [Background] Holzer PW, Leonard DA, Shanmugarajah K, Moulton KN, Ng ZY, Cetrulo CL Jr, Sachs DH. A Comparative Examination of the Clinical Outcome and Histological Appearance of Cryopreserved and Fresh Split-Thickness Skin Grafts. J Burn Care Res. 2017 Jan/Feb;38(1):e55-e61. doi: 10.1097/BCR.0000000000000431. PMID 27606556
- [Derived] Wu D, Zhao XS, Zhao HF, Xie JH, Wei HJ, Zhu NW. New Hope for the Treatment of Severe Skin Injury: Genetically Engineered Porcine Skin Xenotransplantation. Xenotransplantation. 2025 May-Jun;32(3):e70057. doi: 10.1111/xen.70057. PMID 40407357